CLINICAL TRIAL: NCT07292818
Title: Feasibility Study of Novel Applications of Hyaluronic Acid-based Gel Spacers in Gynecologic Malignancies
Brief Title: Hyaluronic Acid-based Gel Spacers in Gynecologic Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Teleflex (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LCCC2310
Record Dates: First submitted 2025-11-24; First posted 2025-12-18 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Cervix Cancer
Keywords: radiotherapy; brachytherapy; gel spacer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Brachytherapy with hyaluronic acid-based gel spacer (Experimental): Patients with cervical cancer who are scheduled to undergo definitive chemoradiotherapy, including brachytherapy, with the use of hyaluronic acid-based gel spacer to increase the distance between the cervix and the anterior rectal wall.
  Interventions: Device: Barrigel gel spacer

INTERVENTIONS:
Device: Barrigel gel spacer — Barrigel (Hyaluronic acid- based gel spacer) will be used to increase the distance between the cervix and the anterior rectal wall, with the intent to decrease the radiation dose delivered to the rectum.
  Other Names: Hyaluronic acid- based rectal spacer

SUMMARY:
This pilot feasibility study evaluates the use of a hyaluronic acid-based spacing gel (Barrigel) in participants with cervical cancer undergoing chemoradiotherapy (chemoRT), including brachytherapy, as part of standard care.

The primary goal is to assess feasibility. Other goals include determining whether gel placement can reduce radiation dose to nearby healthy organs (organs at risk, OAR) and improve delivery of the prescribed radiation dose to the tumor.

In cervical cancer, the radiation dose to the tumor is often limited by the risk of exposing nearby sensitive organs, such as the rectum, bladder, and other pelvic structures. Vaginal packing techniques and specialized devices are used to protect these organs and ensure effective treatment. Gel spacers are inserted before radiation therapy to create space between the rectum and the cervix, reducing radiation exposure to healthy tissue. Already widely used in prostate cancer treatment in the U.S., gel spacers may also help improve tumor control and reduce treatment-related toxicity in cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained to participate in the study and HIPAA authorization for release of personal health information.
* Subject is willing and able to comply with study procedures based on the judgment of the investigator.
* Age ≥ 18 years at time of consent.
* Eastern Cooperative Oncology Group Performance Status of 0-2 or Karnofsky Performance Scale score of 50-100.
* Histological or cytological evidence of cervical cancer. Only patients with cervical cancer who are planned for chemoradiotherapy with brachytherapy, except for individuals with known rectal invasion.

Exclusion Criteria:

* Active infection requiring systemic therapy.
* Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated in the study).
* Known allergy to hyaluronic acid-based products.
* Known inflammatory bowel disease, such as Crohn's disease or ulcerative colitis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cervical carcinoma is seen only in women.
Enrollment: 14 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2030-10-30 (Estimated)

PRIMARY OUTCOMES:
Safety based on Grade 3 or higher adverse events associated with hyaluronic acid-based rectal spacer placement | Up to 3 months after completion of radiotherapy
  The NCI Common Terminology Criteria for Adverse Events (NCI-CTCAE) is a descriptive terminology that can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE. Number of participants with Grade 3 or higher adverse events associated with hyaluronic acid-based rectal spacer placement will be presented.
Safety based on Patient Reported Outcome Report based on The Expanded Prostate Cancer Index Composite (EPIC) Bowel Assessment | Up to 3 months after completion of radiotherapy
  Patient assessments of symptom characteristics will be surveyed based on the Patient Reported Outcome Report, based on the Expanded Prostate Cancer Index Composite (EPIC) Bowel Assessment. Each item in the EPIC bowel domain uses a 5-point Likert scale. The responses are numerically coded and then converted to a 0-100 scale, where higher scores = better function / less bother. No problem=1, very small problem =2, small problem=3, moderate problem=4, big problem=5
Safety based on Patient Reported Outcome Report based on Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Up to 3 months after completion of radiotherapy
  The PRO-CTCAE survey, focused on gastrointestinal and genitourinary symptoms, will be used assessment of toxicity. The PRO-CTCAE Measurement System characterizes the frequency, severity, interference, and presence/absence of symptomatic toxicities reported from the patient perspective. PRO-CTCAE uses 5-point Likert scales to assess the frequency, severity, and daily life interference of patient-reported symptoms, with higher scores indicating more frequent, severe, or bothersome experiences.
Distance between uterus/cervix/proximal vagina and rectum | Up to 7 weeks (at the end of radiotherapy)
  The distance between the uterus, cervix, proximal vagina, and rectum will be measured using images acquired during brachytherapy.
Gel placement procedure time | Up to 7 weeks (at the end of radiotherapy)
  Time required to complete gel placement will be reported.
Difficulty of gel placement | Up to 7 weeks (at the end of radiotherapy)
  Difficulty of Barrigel Procedure Insertion will be graded based on provider response to a 4-point scale survey. Higher scores represent difficult insertions. 1- Very Easy: All anatomical landmarks were easy to spot on transrectal ultrasonogram (TRUS), and Barrigel was well-visualized during injection. The tissue is separated well with Barrigel. Visible spacing between the cervix and rectum was achieved. The implant was positioned well and sculpted to the desired (symmetric) shape. 2- Easy: Most landmarks were easily seen, Barrigel was well-visualized, tissue separated reasonably well overall, although the shape may not be ideal. 3- Difficult: Some anatomy or Barrigel was difficult to visualize on TRUS, and/or the tissue didn't separate well in places with Barrigel. Spacing goals were notably not achieved, but some useful space was provided. 4- Very Difficult: The TRUS visibility was compromised, and/or the gel didn't get injected as planned due to tissue.

SECONDARY OUTCOMES:
Implant geometry | Up to 7 weeks (at the end of radiotherapy)
  Implant geometry will be characterized using a T2-weighted magnetic resonance imaging (MRI). The anatomic location of the implant will be specified qualitatively. Measurements obtained will include maximum length, width, and thickness of implant overall. Descriptive statistics (mean/sd) for measurements of implant geometry will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Shivani Sud, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials